CLINICAL TRIAL: NCT05984784
Title: A Phase1b/2a Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of IMG-007 in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of IMG-007 in Adults With Atopic Dermatitis (AD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Cohort 1 was completed. Cohort 2 was cancelled because data from Cohort 1 provided sufficient information for further development decision. No safety concerns were noted.
Sponsor: Inmagene LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMG-007-201
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis; Moderate-to-severe Atopic Dermatitis; AD
Keywords: IMG-007; Atopic Dermatitis; Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Immune System Diseases; Dermatologic Agents
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 IMG-007 Dose 1 (Experimental): IMG-007 Dose 1 will be administered intravenously 3 times over 4 weeks
  Interventions: Drug: IMG-007
- Cohort 2 IMG-007 Dose 2 (Experimental): IMG-007 Dose 2 will be administered intravenously 3 times over 4 weeks
  Interventions: Drug: IMG-007
- Placebo (Placebo Comparator): Placebo will be administered intravenously 3 times over 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Drug: Placebo Intravenous Infusion
  Arms: Placebo
Drug: IMG-007 — Drug: IMG-007 Intravenous Infusion
  Arms: Cohort 1 IMG-007 Dose 1; Cohort 2 IMG-007 Dose 2

SUMMARY:
The primary objective of this study is to evaluate the safety of IMG-007 in adults with moderate-to-severe AD. The secondary objectives are to evaluate the pharmacokinetics and efficacy of IMG-007 in AD patients.

DETAILED DESCRIPTION:
This is a phase 1b/2a study to assess the safety, tolerability, PK, efficacy, and PD of multiple doses of IMG-007 in participants with AD. The study will consist of two cohorts with three periods: a screening period of up to 5 weeks, a 12-week treatment period, and a 12-week follow-up period. Cohort 1 is open-label, with approximately 15 participants to receive three IV infusions of IMG-007 Dose 1 over 4 weeks. Cohort 2 is randomized, double-blind and placebo-controlled, with approximately 40 participants to be randomized in a 3:1 ratio to receive three IV infusions of IMG-007 Dose 2 or matching placebo over 4 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged ≥ 18 and < 75 years.
* Moderate-to-severe AD.
* Documented history of inadequate response or lack of tolerability to a stable regimen of one or more topical treatment before the Screening visit, or for whom topical treatments are otherwise inadvisable.
* Female participants who are not pregnant or breastfeeding and meet at least one of the following conditions: not of childbearing potential or of childbearing potential and agrees to use a highly effective method of contraception.

Key Exclusion Criteria:

* Known hepatitis B, hepatitis C, or human immunodeficiency virus infection.
* Evidence of active or latent tuberculosis (TB).
* History of untreated or inadequately treated TB infection.
* Active infection requiring treatment with systemic antibiotics, antivirals, antifungals, antiparasitics or antiprotozoals at the Screening visit.
* Active unstable pruritic skin conditions in addition to AD that would interfere with the assessment of AD based on the investigator's clinical judgement.
* Other conditions or laboratory abnormality that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - Amicis Research Center, Northridge, California
  - Amicis Research Center, Valencia, California
  - Medical Research Center of Miami II Inc, Miami, Florida
  - Optimal Research Sites, Orange City, Florida
  - USF Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida
  - Revival Research Institute, LLC, Troy, Michigan
  - Markowitz Medical, LLC, New York, New York
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
- Canada (3):
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - DermEffects, London, Ontario
  - Centre de Recherche Saint-Louis (Québec), Québec

IPD SHARING:
Plan to Share IPD: Undecided
Data to be disclosed for primary and secondary endpoints.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 IMG-007 Dose 1: IMG-007 Dose 1 was to be administered intravenously 3 times over 4 weeks
  IMG-007: Drug: IMG-007 Intravenous Infusion
Period: Overall Study
Arm/Group | Cohort 1 IMG-007 Dose 1
Started | 13
Completed | 8
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1 IMG-007 Dose 1
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
EASI score [Mean (Standard Deviation); unit: units on a scale] — The eczema area and severity index (EASI) is a validated composite scoring system assessed by the investigator based on the body area involved in each of the four body regions (head and neck, upper limbs, lower limbs, and trunk) and the average severity of each of the four key signs of AD (erythema, edema/papulation, excoriation, and lichenification) based on a 4-point scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The total EASI score ranges from 0 (clear or no eczema) to 72 (maximum severity), with higher values indicating more severe and/or extensive disease.
  units on a scale | 29.5 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Adverse Events in Participants
Description: To evaluate adverse events (AEs) emergent from multiple doses of IMG-007 in adult participants with atopic dermatitis (AD)
Time Frame: Adverse events were collected from baseline through the end of the study, a period of up to 24 weeks.
Measure: Number; unit: participants
Arm/Group | Cohort 1 IMG-007 Dose 1
Number analyzed (Participants) | 13
participants
  Participants with at least 1 TEAE | 9
  SAE | 0
  Investigational product-related TEAE | 0
  TEAE that was an infusion-related reaction | 0
  TEAE leading to 4-week dosing period discontinuation | 0
  TEAE with outcome of death | 0

2. Secondary Outcome: Pharmacokinetic Characterization
Description: To characterize the pharmacokinetic (PK) profile of multiple doses of IMG-007 in AD participants
Time Frame: Serum concentrations of IMG-007 were measured at Week 4 (pre-dose and post-dose), Week 12 (post-dose), and Week 24 (post-dose).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 IMG-007 Dose 1
Number analyzed (Participants) | 13
ng/mL
  Week 4, Pre-dose | 47650.0 (16255.6)
  Week 4, Post-dose | 131400.0 (18379.3)
  Week 12, Post-dose | 16088.0 (12662.2)
  Week 24, Post-Dose | 1334.2 (1720.5)

3. Secondary Outcome: Evaluation of Eczema Area and Severity Index (EASI)
Description: The Eczema Area and Severity Index (EASI) is a validated composite scoring system assessed by the investigator based on the body area involved in each of the four body regions (head and neck, upper limbs, lower limbs, and trunk) and the average severity of each of the four key signs of AD (erythema, edema/papulation, excoriation, and lichenification) based on a 4-point scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The total EASI score ranges from 0 (clear or no eczema) to 72 (maximum severity), with higher values indicating more severe and/or extensive disease.
Time Frame: Mean percent change from baseline in Eczema Area and Severity Index (EASI) at week 12.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Cohort 1 IMG-007 Dose 1
Number analyzed (Participants) | 13
percentage of change | -68.5 (11.4)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Cohort 1 IMG-007 Dose 1
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 IMG-007 Dose 1 (N=13)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2
COVID-19 (Infections and infestations) | 1
localized infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT05984784/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT05984784/SAP_001.pdf